CLINICAL TRIAL: NCT01840657
Title: Prospective Study of Adverse Event Rates in Males With X-Linked Myotubular Myopathy
Brief Title: Myotubular Myopathy Event Study
Acronym: MTMES
Status: Completed | Type: Observational
Sponsor: Cure CMD (Other)
Collaborators: Congenital Muscle Disease International Registr (Other); University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: CMDIR-002
Record Dates: First submitted 2013-04-18; First posted 2013-04-26 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2017-01

CONDITIONS: X-linked Myotubular Myopathy
Keywords: CMDIR (Congenital Muscle Disease International Registry); X-linked myotubular myopathy; centronuclear myopathy; myotubularin; MTM1 gene; mutation; survival; adverse event; disease complication; hospital admission; emergency room visit; motor function; respiratory function; natural history study
MeSH Terms: conditions — Myopathies, Structural, Congenital; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
X-Linked myotubular myopathy (XLMTM), a form of centronuclear myopathy (CNM) is the result of a mutation in the MTM1 (myotubularin) gene which leads to altered myotubularin. Myotubularin is essential for optimum muscle function. To date, over 100 mutations have been described resulting in a range of disease onset and symptom severity. The early onset form presents with neonatal hypotonia, muscle weakness, respiratory distress and an ongoing requirement for continuous ventilatory support with the inability to maintain a sitting position once placed. Males with both later onset and milder symptoms usually do not require ongoing ventilatory support, achieve a higher maximal motor function with ability to sit when placed and even walk, and have improved survival rates. Males with XLMTM may experience complications (events) at birth and throughout their lifetime. The goal of the study is to identify the number of events over twelve months in males with genetically confirmed XLMTM. Parents or affected individuals over the age of 18 years who are able to access telephone will provide answers to an established event survey to evaluate the frequency and types of events. Emergency department, hospital admissions and mortality will be confirmed by obtaining medical reports.

The investigators hypothesize that there will be no association between the frequency of events and markers of clinical severity including the need for ventilatory support at birth, current level of ventilatory support (no support, support less than 12 hours, support more than 12 hours) and current motor function (walking, sitting without support, inability to sit without support).

ELIGIBILITY:
Inclusion Criteria:

* males with a confirmed MTM1 mutation OR
* males with a muscle biopsy consistent with myotubular myopathy AND family history consistent with X-linked inheritance AND
* English-speaking parent/guardian of a living male child or a decisionally impaired adult OR English-speaking affected male over 18 years of age who can access telephone
* signed study consent
* enrolled in the Congenital Muscle Disease International Registry (CMDIR)

Exclusion Criteria:

* males with only a clinical diagnosis of XLMTM but without family history of XLMTM
* an affected male who has a genetically confirmed form of centronuclear myopathy (CNM) that is not caused by a mutation in the MTM1 gene
* females with MTM1 due to the limited number of females affected and the variability of clinical presentation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants for the MTM Event study will be recruited from 2 sources:
  * the Centronculear Myopathy Natural History Study and
  * the Congenital Muscle Disease International Registry (CMDIR)
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Survey of a defined set of events | 12 months
  Changes in care needed, breathing support, motor ability, medications and medical care, nutrition/weight management, communication/vision/learning/behavior, and frequency of outpatient/hospital/ER visits are recorded by a monthly telephone survey.
Frequency of a predefined set of events related to ventilatory status | 12 months
  To analyze the strength of the association between the frequency of events surveyed and 1) duration of ventilatory support directly after birth and 2) current need for ventilatory support.
Frequency of a predefined set of events related to current motor function | 12 months
  To analyze the strength of the association between the frequency of events surveyed and current motor function

SECONDARY OUTCOMES:
Association between event frequency and genotype | 12 months
  To determine the strength of the association between the frequency of the events surveyed and the affected individual's genotype.
Association between event rate and season | 12 months
  To analyze event rates with respect to two seasonal clusters, October through March and April through September.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hornyak, MD, PhD, Principal Investigator — University of Michigan; Anne Rutkowski, MD, Principal Investigator — Cure CMD; James Dowling, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- CMDIR, Torrance, California, United States

REFERENCES:
- [Background] Al-Qusairi L, Laporte J. T-tubule biogenesis and triad formation in skeletal muscle and implication in human diseases. Skelet Muscle. 2011 Jul 13;1(1):26. doi: 10.1186/2044-5040-1-26. PMID 21797990
- [Background] Al-Qusairi L, Weiss N, Toussaint A, Berbey C, Messaddeq N, Kretz C, Sanoudou D, Beggs AH, Allard B, Mandel JL, Laporte J, Jacquemond V, Buj-Bello A. T-tubule disorganization and defective excitation-contraction coupling in muscle fibers lacking myotubularin lipid phosphatase. Proc Natl Acad Sci U S A. 2009 Nov 3;106(44):18763-8. doi: 10.1073/pnas.0900705106. Epub 2009 Oct 21. PMID 19846786
- [Background] Beggs AH, Bohm J, Snead E, Kozlowski M, Maurer M, Minor K, Childers MK, Taylor SM, Hitte C, Mickelson JR, Guo LT, Mizisin AP, Buj-Bello A, Tiret L, Laporte J, Shelton GD. MTM1 mutation associated with X-linked myotubular myopathy in Labrador Retrievers. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14697-702. doi: 10.1073/pnas.1003677107. Epub 2010 Aug 3. PMID 20682747
- [Background] Biancalana V, Caron O, Gallati S, Baas F, Kress W, Novelli G, D'Apice MR, Lagier-Tourenne C, Buj-Bello A, Romero NB, Mandel JL. Characterisation of mutations in 77 patients with X-linked myotubular myopathy, including a family with a very mild phenotype. Hum Genet. 2003 Feb;112(2):135-42. doi: 10.1007/s00439-002-0869-1. Epub 2002 Nov 28. PMID 12522554
- [Background] Buj-Bello A, Biancalana V, Moutou C, Laporte J, Mandel JL. Identification of novel mutations in the MTM1 gene causing severe and mild forms of X-linked myotubular myopathy. Hum Mutat. 1999;14(4):320-5. doi: 10.1002/(SICI)1098-1004(199910)14:43.0.CO;2-O. PMID 10502779
- [Background] Buj-Bello A, Fougerousse F, Schwab Y, Messaddeq N, Spehner D, Pierson CR, Durand M, Kretz C, Danos O, Douar AM, Beggs AH, Schultz P, Montus M, Denefle P, Mandel JL. AAV-mediated intramuscular delivery of myotubularin corrects the myotubular myopathy phenotype in targeted murine muscle and suggests a function in plasma membrane homeostasis. Hum Mol Genet. 2008 Jul 15;17(14):2132-43. doi: 10.1093/hmg/ddn112. Epub 2008 Apr 22. PMID 18434328
- [Background] Cao C, Backer JM, Laporte J, Bedrick EJ, Wandinger-Ness A. Sequential actions of myotubularin lipid phosphatases regulate endosomal PI(3)P and growth factor receptor trafficking. Mol Biol Cell. 2008 Aug;19(8):3334-46. doi: 10.1091/mbc.e08-04-0367. Epub 2008 Jun 4. PMID 18524850
- [Background] Dowling JJ, Lawlor MW, Das S. X-Linked Myotubular Myopathy. 2002 Feb 25 [updated 2018 Aug 23]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1432/ PMID 20301605
- [Background] de Gouyon BM, Zhao W, Laporte J, Mandel JL, Metzenberg A, Herman GE. Characterization of mutations in the myotubularin gene in twenty six patients with X-linked myotubular myopathy. Hum Mol Genet. 1997 Sep;6(9):1499-504. doi: 10.1093/hmg/6.9.1499. PMID 9285787
- [Background] Dowling JJ, Gibbs EM, Feldman EL. Membrane traffic and muscle: lessons from human disease. Traffic. 2008 Jul;9(7):1035-43. doi: 10.1111/j.1600-0854.2008.00716.x. Epub 2008 Feb 4. PMID 18266915
- [Background] Dowling JJ, Vreede AP, Low SE, Gibbs EM, Kuwada JY, Bonnemann CG, Feldman EL. Loss of myotubularin function results in T-tubule disorganization in zebrafish and human myotubular myopathy. PLoS Genet. 2009 Feb;5(2):e1000372. doi: 10.1371/journal.pgen.1000372. Epub 2009 Feb 6. PMID 19197364
- [Background] Herman GE, Finegold M, Zhao W, de Gouyon B, Metzenberg A. Medical complications in long-term survivors with X-linked myotubular myopathy. J Pediatr. 1999 Feb;134(2):206-14. doi: 10.1016/s0022-3476(99)70417-8. PMID 9931531
- [Background] Herman GE, Kopacz K, Zhao W, Mills PL, Metzenberg A, Das S. Characterization of mutations in fifty North American patients with X-linked myotubular myopathy. Hum Mutat. 2002 Feb;19(2):114-21. doi: 10.1002/humu.10033. PMID 11793470
- [Background] Hoffjan S, Thiels C, Vorgerd M, Neuen-Jacob E, Epplen JT, Kress W. Extreme phenotypic variability in a German family with X-linked myotubular myopathy associated with E404K mutation in MTM1. Neuromuscul Disord. 2006 Nov;16(11):749-53. doi: 10.1016/j.nmd.2006.07.020. Epub 2006 Sep 26. PMID 17005396
- [Background] Joseph M, Pai GS, Holden KR, Herman G. X-linked myotubular myopathy: clinical observations in ten additional cases. Am J Med Genet. 1995 Nov 6;59(2):168-73. doi: 10.1002/ajmg.1320590211. PMID 8588581
- [Background] Jungbluth H, Wallgren-Pettersson C, Laporte J. Centronuclear (myotubular) myopathy. Orphanet J Rare Dis. 2008 Sep 25;3:26. doi: 10.1186/1750-1172-3-26. PMID 18817572
- [Background] Laporte J, Biancalana V, Tanner SM, Kress W, Schneider V, Wallgren-Pettersson C, Herger F, Buj-Bello A, Blondeau F, Liechti-Gallati S, Mandel JL. MTM1 mutations in X-linked myotubular myopathy. Hum Mutat. 2000;15(5):393-409. doi: 10.1002/(SICI)1098-1004(200005)15:53.0.CO;2-R. PMID 10790201
- [Background] Lee IC, Su PH, Chen JY, Hu JM, Lu JJ, Ng YY. Congenital myotubular myopathy with a novel MTM1 gene mutation in a premature infant presenting with ventilator dependency and intrahepatic cholestasis. J Child Neurol. 2012 Jan;27(1):99-104. doi: 10.1177/0883073811414419. Epub 2011 Aug 31. PMID 21881007
- [Background] Penisson-Besnier I, Biancalana V, Reynier P, Cossee M, Dubas F. Diagnosis of myotubular myopathy in the oldest known manifesting female carrier: a clinical and genetic study. Neuromuscul Disord. 2007 Feb;17(2):180-5. doi: 10.1016/j.nmd.2006.10.008. Epub 2007 Jan 23. PMID 17251023
- [Background] Romero NB, Bitoun M. Centronuclear myopathies. Semin Pediatr Neurol. 2011 Dec;18(4):250-6. doi: 10.1016/j.spen.2011.10.006. No abstract available. PMID 22172420
- [Background] Robinson FL, Dixon JE. Myotubularin phosphatases: policing 3-phosphoinositides. Trends Cell Biol. 2006 Aug;16(8):403-12. doi: 10.1016/j.tcb.2006.06.001. Epub 2006 Jul 7. PMID 16828287